CLINICAL TRIAL: NCT05098132
Title: A Phase 1/2 Study to Evaluate STK-012 as a Single Agent and in Combination Therapy in Subjects With Front-line Advanced NSCLC and Other Selected Indications
Brief Title: Study of STK-012 Alone and With Other Treatments in Patients With Advanced Lung Cancer and Other Cancers
Acronym: SYNERGY-101
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Synthekine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STK-012-101
Record Dates: First submitted 2021-10-06; First posted 2021-10-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor; Non Small Cell Lung Cancer; Untreated Advanced NSCLC; 1st Line NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Phase 1a: STK-012 monotherapy dose escalation (Experimental): STK-012 subcutaneous (SC) as monotherapy in selected solid tumor indications
  Interventions: Drug: STK-012
- Phase 1a: STK-012 + pembrolizumab dose escalation (Experimental): STK-012 SC + pembrolizumab intravenously (IV) in selected solid tumor indications
  Interventions: Drug: STK-012; Drug: pembrolizumab
- Phase 1a: STK-012 + standard of care (SoC) dose escalation (Experimental): STK-012 SC + SoC IV in first-line non-squamous (NSQ) NSCLC
  Interventions: Drug: STK-012; Drug: pembrolizumab; Drug: pemetrexed; Drug: carboplatin
- Phase 1b: STK-012 monotherapy expansion (Experimental): STK-012 SC monotherapy in selected solid tumor indications
  Interventions: Drug: STK-012
- Phase 1b: STK-012 + pembrolizumab dose expansion (Experimental): STK-012 SC will be administered in combination with pembrolizumab IV in selected solid tumor indications
  Interventions: Drug: STK-012; Drug: pembrolizumab
- Phase 1b: STK-012 + SoC dose expansion (Experimental): STK-012 SC + SoC IV in first-line PD-L1 negative NSQ NSCLC
  Interventions: Drug: STK-012; Drug: pembrolizumab; Drug: pemetrexed; Drug: carboplatin
- Phase 2: Arm A (Experimental): STK-012 2.25 mg SC Q3W + SoC IV in first-line PD-L1 negative NSQ NSCLC
  Interventions: Drug: STK-012; Drug: pembrolizumab; Drug: pemetrexed; Drug: carboplatin
- Phase 2: Arm B (Experimental): STK-012 1.5 mg SC Q3W + SoC IV in first-line PD-L1 negative NSQ NSCLC
  Interventions: Drug: STK-012; Drug: pembrolizumab; Drug: pemetrexed; Drug: carboplatin
- Phase 2: Arm C (Active Comparator): SoC IV in first-line PD-L1 negative NSQ NSCLC
  Interventions: Drug: pembrolizumab; Drug: pemetrexed; Drug: carboplatin

INTERVENTIONS:
Drug: STK-012 — Engineered Interleukin-2 (IL-2) selective for antigen activated T cells
  Arms: Phase 1a: STK-012 + pembrolizumab dose escalation; Phase 1a: STK-012 + standard of care (SoC) dose escalation; Phase 1a: STK-012 monotherapy dose escalation; Phase 1b: STK-012 + SoC dose expansion; Phase 1b: STK-012 + pembrolizumab dose expansion; Phase 1b: STK-012 monotherapy expansion; Phase 2: Arm A; Phase 2: Arm B
Drug: pembrolizumab — anti-PD-1 monoclonal antibody
  Arms: Phase 1a: STK-012 + pembrolizumab dose escalation; Phase 1a: STK-012 + standard of care (SoC) dose escalation; Phase 1b: STK-012 + SoC dose expansion; Phase 1b: STK-012 + pembrolizumab dose expansion; Phase 2: Arm A; Phase 2: Arm B; Phase 2: Arm C
Drug: pemetrexed — chemotherapy
  Arms: Phase 1a: STK-012 + standard of care (SoC) dose escalation; Phase 1b: STK-012 + SoC dose expansion; Phase 2: Arm A; Phase 2: Arm B; Phase 2: Arm C
Drug: carboplatin — chemotherapy
  Arms: Phase 1a: STK-012 + standard of care (SoC) dose escalation; Phase 1b: STK-012 + SoC dose expansion; Phase 2: Arm A; Phase 2: Arm B; Phase 2: Arm C

SUMMARY:
This is a phase 1/2, multicenter, open-label study. The phase 1 portion is a dose escalation and expansion study of STK-012 as monotherapy and in combination therapy in patients with selected advanced solid tumors. The phase 2 portion is a randomized study of STK-012 in combination with standard of care (SoC) pembrolizumab, pemetrexed, and carboplatin versus SoC, in patients with first line, PD-L1 negative, non-squamous, non-small cell lung cancer.

DETAILED DESCRIPTION:
Phase 1 [closed to enrollment]: The phase 1a portion is a dose escalation study to evaluate STK-012 as monotherapy and in combination therapy in patients with selected solid tumors. The phase 1b portion is a dose expansion study to evaluate STK-012 as monotherapy and in combination therapy at the candidate recommended phase 2 dose (RP2D) in selected solid tumor types.

Phase 2 [open to enrollment]: The phase 2 portion is a randomized, open label study to evaluate STK-012 at two dose levels in combination with standard of care (SoC) pembrolizumab, pemetrexed and carboplatin, versus SoC, in patients with first line, PD-L1 negative, non-squamous, non-small cell lung cancer.

ELIGIBILITY:
Selected Inclusion Criteria:

1. Phase 1 [closed to enrollment]
2. Phase 2 [open to enrollment]:

   * Diagnosis of non-small cell lung cancer (NSCLC).
   * Stage IV or Stage IIIB/IIIC and not a candidate for definitive treatment.
   * Non-squamous (NSQ) cell histology.
   * No prior systemic therapy for advanced/metastatic NSQ NSCLC.
   * Tumor is PD-L1 negative (TPS <1%) by local testing.
   * No known actionable EGFR, ALK, ROS1, or other actionable genomic aberrations for which there is a local standard of care available as front line therapy.

Selected Exclusion Criteria:

1. Phase 1 [closed to enrollment]
2. Phase 2 [open to enrollment]:

   * Prior immune checkpoint inhibitor (anti-PD[L]1 and/or anti-CTLA-4) treatment
   * Tumor with small cell, neuroendocrine, or sarcomatoid components.
   * Received radiotherapy ≤ 7 days of the first dose of study treatment.
   * Known untreated central nervous system metastases
   * Any history of carcinomatous meningitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Treatment emergent adverse events (TEAEs) | From 1st dose of study treatment through 90 days after last dose
  Incidence of TEAEs in participants with select advanced solid tumors
Phase 1a: Serious adverse events (SAEs) | From 1st dose of study treatment through 90 days after last dose
  Incidence of SAEs in participants with select advanced solid tumors
Phase 1a: Dose limiting toxicities (DLTs) | Cycle 1, Days 1 through 21
  Incidence of DLTs in participants with select advanced solid tumors
Phase 1a: Deaths | From 1st dose of study treatment until death, up to 4 years
  Incidence of death in participants with select advanced solid tumors
Phase 1b: TEAEs at the RP2D | From 1st dose of study treatment through 90 days after last dose
  Incidence of TEAEs at the recommended phase 2 dose (RP2D) in participants with select advanced solid tumors
Phase 1b: SAEs at the RP2D | From 1st dose of study treatment through 90 days after last dose
  Incidence of SAEs at the RP2D in participants with select advanced solid tumors
Phase 1b: Deaths at the RP2D | From 1st dose of study treatment until death, up to 4 years
  Incidence of death at the RP2D in participants with select advanced solid tumors
Phase 2: Overall response rate (ORR) in Arm A versus Arm C | From randomization until disease progression or death, or the last evaluable assessment in the absence of progression, up to 4 years
  To compare the ORR in 1L PD-L1 negative NSQ NSCLC subjects treated with STK-012 2.25 mg + SoC vs. SoC (Arms A vs. C). ORR is the proportion of subjects with confirmed complete response (CR) or confirmed partial response (PR) per BICR.

SECONDARY OUTCOMES:
Phase 1: ORR | From enrollment until disease progression or death, or the last evaluable assessment in the absence of progression, up to 4 years
  Assessment of preliminary efficacy, specifically ORR, in select advanced solid tumors. ORR is the proportion of subjects with confirmed CR or confirmed PR per investigator assessment.
Phase 1: Progression free survival (PFS) | From enrollment until first documentation of disease progression per investigator assessment or death due to any cause, whichever occurs first, up to 4 years
  Assessment of preliminary efficacy, specifically PFS, in select advanced solid tumors.
Phase 1: Overall survival (OS) | From enrollment until death due to any cause, up to 4 years
  Assessment of preliminary efficacy, specifically OS, in select advanced solid tumors.
Phase 1/2: STK-012 ADAs | From screening through 30 days after last dose of STK-012
  Anti-drug antibodies (ADA) to assess immunogenicity of STK-012 in advanced NSCLC and other select solid tumors.
Phase 1/2: AUC of STK-012 | From screening through 30 days after last dose of STK-012
  Area under the curve (AUC) to assess pharmacokinetic (PK) characterization of STK-012 in advanced NSCLC and other select solid tumors.
Phase 1/2: Cmax of STK-012 | From screening through 30 days after last dose of STK-012
  Maximum concentration (Cmax) to assess PK characterization of STK-012 in advanced NSCLC and other select solid tumors.
Phase 1/2: Tmax of STK-012 | From screening through 30 days after last dose of STK-012
  Time of maximum concentration (Tmax) to assess PK characterization of STK-012 in advanced NSCLC and other select solid tumors.
Phase 1/2: Half life of STK-012 | From screening through 30 days after last dose of STK-012
  Half life (t1/2) to assess PK characterization of STK-012 in advanced NSCLC and other select solid tumors.
Phase 2: PFS in Arm A versus Arm C | From randomization until first documentation of disease progression per BICR or death due to any cause, whichever occurs first, up to 4 years
  To compare the PFS in 1L PD-L1 negative NSQ NSCLC subjects treated with STK-012 2.25 mg + SoC vs. SoC (Arms A vs. C). PFS is the time from randomization until the first documentation of disease progression per BICR or death due to any cause, whichever occurs first.
Phase 2: ORR in Arm B versus Arm C | From randomization until disease progression or death, or the last evaluable assessment in the absence of progression, up to 4 years
  To compare the ORR in 1L PD-L1 negative NSQ NSCLC subjects treated with STK-012 1.5 mg + SoC vs. SoC (Arms B vs. C). ORR is the proportion of subjects with confirmed CR or confirmed PR per BICR.
Phase 2: PFS in Arm B versus Arm C | From randomization until first documentation of disease progression per BICR or death due to any cause, whichever occurs first, up to 4 years
  To compare the PFS in 1L PD-L1 negative NSQ NSCLC subjects treated with STK-012 1.5 mg + SoC vs. SoC (Arms B vs. C). PFS is the time from randomization until the first documentation of disease progression per BICR or death due to any cause, whichever occurs first.
Phase 2: OS in Arm A versus C | From randomization until death due to any cause, up to 4 years
  To compare the OS in 1L PD-L1 negative NSQ NSCLC subjects treated with STK-012 2.25 mg + SoC vs. SoC (Arms A vs. C). OS is the time from randomization until death due to any cause.
Phase 2: OS in Arm B versus C | From randomization until death due to any cause, up to 4 years
  To compare the OS in 1L PD-L1 negative NSQ NSCLC subjects treated with STK-012 1.5 mg + SoC vs. SoC (Arms B vs. C). OS is the time from randomization until death due to any cause.
Phase 2: TEAEs | From 1st dose of study treatment through 90 days after last dose
  Incidence of TEAEs in 1L PD-L1 negative NSQ NSCLC
Phase 2: SAEs | From 1st dose of study treatment through 90 days after last dose
  Incidence of SAEs in 1L PD-L1 negative NSQ NSCLC
Phase 2: Deaths | From 1st dose of study treatment until death, up to 4 years
  Incidence of death in 1L PD-L1 negative NSQ NSCLC

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Providence Medical Foundation, Fullerton, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - Yale New Haven Hospital, Yale Cancer Center, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - HealthPartners Cancer Center at Regions Hospital, Saint Paul, Minnesota
  - Northwell Health, Lake Success, New York
  - NYU Langone Health, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Baptist Memorial Hospital Cancer Center, Memphis, Tennessee
  - Sarah Cannon Research Institute - Nashville, Nashville, Tennessee
  - Renovatio Clinical, El Paso, Texas
  - Oncology Consultants, Houston, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - NEXT Virginia, Fairfax, Virginia
  - Northwest Medical Specialties, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No